CLINICAL TRIAL: NCT05102305
Title: A Multi-center, Prospective, Observational Study to Evaluate the Effectiveness of N-acetylcysteine (NAC) Nebulizer Therapy (Mucomyst Solution) in COPD With Difficulty of Expectoration
Brief Title: A Multi-center,Prospective, OS to Evaluate the Effectiveness of 'NAC' Nebulizer Therapy in COPD (NEWEST)
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-NAC-OS-402
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the effect of Mucomyst nebulizer therapy on improvement in symptoms and quality of life in COPD patients with difficulty of expectoration.

DETAILED DESCRIPTION:
In this non-interventional observational study, treatment for individual subjects is determined by the investigator according to the status of individual subjects in routine clinical practice. In this circumstance, doses for each drug product will not be specified in the protocol but will be determined as appropriate by the investigator with the product label and the subject's medical condition taken into consideration.

Primary objective To evaluate the effect of Mucomyst on improvement in difficulty of expectoration symptoms in COPD patients with difficulty of expectoration.

Secondary objective To evaluate the effect of Mucomyst on improvement in quality of life and safety in COPD patients with difficulty of expectoration.

ELIGIBILITY:
Inclusion Criteria:

1. man and woman at the age of ≥40 years old
2. Diagnosed with COPD within the past 1 year based on pulmonary function test (post bronchodilator FEV1/FVC<0.7)
3. COPD Assessment Test (CAT) phlegm score ≥2
4. Smoking history ≥10 pack-years* (*Pack-year: number of packs of cigarettes smoked per day X number of years the individual has smoked)
5. Patient who is to be treated with Mucomyst nebulizer therapy to alleviate difficulty of expectoration symptoms
6. Voluntary written informed consent to study participation and to use of personal information for this study

Exclusion criteria

1. History of hypersensitivity reactions to any of the components of NAC or contraindicated to NAC therapy according to the product label
2. Treated with Mucomyst within the past 4 weeks
3. Newly treated with 'drugs for the alleviation of expectoration symptoms (antitussives/expectorants)' or dose changed for ongoing therapy within the past 4 weeks
4. Pregnant and lactating woman
5. Participating in another trial with investigational product treatment at the time of enrollment to the present study
6. Ineligible for study participation in the opinion of the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease (COPD) patients with Difficulty of Expectoration. Total 100 subjects
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in CAT | at Week 12
  Change from baseline in CAT phlegm score at Week 12

SECONDARY OUTCOMES:
Change from baseline in CAT | at Weeks 4 and 8
  Change from baseline in CAT phlegm score at Weeks 4 and 8
Change from baseline in CAT | at Weeks 4, 8,and 12
  Change from baseline in CAT total score and sub-scale score at Weeks 4, 8, and 12
Change from baseline in SGRQ-C | at Weeks 4, 8, and 12
  Change from baseline in St. George's Respiratory Questionnaire for COPD patients (SGRQ-C) total score at Weeks 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: MyungSook Hong, Study Director — MOG
Locations (1):
- The Konkuk University medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No